CLINICAL TRIAL: NCT06707662
Title: Left Septal Pacing or Left Bundle Branch Pacing to Avoid Left Ventricle Systolic Dysfunction. A Multicenter Randomized Trial From the STAY Investigators
Brief Title: Left Septal Pacing or Left Bundle Branch Pacing to Avoid Left Ventricle Systolic Dysfunction
Acronym: STAY II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Ermengol Vallès, Director of Electrophysiology and Cardiac Stimulation Program, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024/11667/I
Record Dates: First submitted 2024-11-19; First posted 2024-11-27 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: AV Block
Keywords: Conduction System Pacing; Left bundle branch area pacing; Right ventricle apical pacing; Left septum pacing; Left ventricle ejection fraction; Heart failure
MeSH Terms: conditions — Atrioventricular Block; Heart Failure | interventions — Defibrillators

STUDY DESIGN:
Intervention Model Description: The study arm will be defined by randomization immediately before the implantation. Patients randomized to RVAP group will undergo an apex ventricular lead. In patients receiving a LBBAP CSP lead, the procedure will be anatomicaly guided, aiming for a "W" pattern in V1 during septal maping. Operators then will screw the lead, aiming for a moderate drop in the impedance, together with the conversion of the "W" pattern into a qR or rSR pattern in lead V1. The current of injury (COI) will be additionally used as a guide. The cornerstone of this study will be to accept the first location as the final location, as long as unipolar and bipolar thresholds are optimal, and the RBBB pattern in lead V1 remains. To ensure a balanced distribution between LBBP and LVSP, the first operator will not have access to any criteria measurement during the implant procedure, but the morphology in V1. After the procedure investigators will fulfill the Redcap database with all the banned EPRS measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Right Ventricle Apical Pacing (Active Comparator): Standard location for any pacing lead in the right ventricle
  Interventions: Device: Pacemaker and defibrillator
- Left bundle branch pacing (Experimental): Stimulation in the Conduction System (righ ventricle) capturing the left budle branch
  Interventions: Device: Pacemaker and defibrillator
- Left septal pacing (Experimental): Stimulation in the Conduction System (righ ventricle) without capturing the left budle branch
  Interventions: Device: Pacemaker and defibrillator

INTERVENTIONS:
Device: Pacemaker and defibrillator — Pacemaker implantation, which can be a regular right ventricle apical lead or a LBBAP lead (LBBP or LVSP dependint on the criteria accomplished).

SUMMARY:
Right ventricular apical pacing (RVAP) can produce left ventricular dysfunction (LVD). Conduction system pacing (CSP) has been used successfully to reverse LVD in patients with left bundle branch block. A recent randomized controlled trial (RCT) has demonstrated that CSP, mostly performed with left bundle branch area pacing (LBBAP), can preserve normal ventricular function and heart failure admissions compared to RVAP in the setting of a high burden of ventricular pacing11 (Stay Trial).

Criteria to assess the LBBAP distinguishes those cases in which the LBB is captured (LBBP) from those in which only the muscular septum surrounding the LBB is captured (LVSP). To date, data regarding LVSP to preserve left ventricle ejection fraction (LVEF) is scarce and limited to non-randomized studies.

DETAILED DESCRIPTION:
Conventional right ventricular apical pacing (RVAP) can produce electrical and mechanical dysynchrony, which may lead to left ventricle dysfunction (LVD) in up to 12% of patients with normal left ventricle ejection fraction (LVEF). A high burden on RVAP is a major predictor of developing LVD, atrial fibrillation (AF), heart failure (HF), and mortality. CSP is able to preserve a more physiological pattern of cardiac electrical activation, utilizing the native conduction system network, or correcting a bundle branch block morphology in patients with disturbances at a proximal or intermediate level of the conduction system network.

The aim of the study is to demonstrate that LVSP can preserve ventricular function compared to LBBP in patients with preserved or mildly deteriorated LVEF and a high burden of expected ventricular pacing. A second hypothesis is to demonstrate than both LVSP and LBBP are both superior to RVAP.

Study design The STAY II trial is a multi-center, prospective, randomized, parallel, controlled study, comparing 12 months outcomes in a population undergoing pacemaker implantation due to a high degree atrio-ventricular block (AVB). All patients will sign informed consent and will be implanted with a pacemaker in a 1:2 randomized fashion to conventional RVAP vs LBBAP (LBBP or LVSP). Randomization to RVAP or LBBAP will be performed during the pre-procedural antibiotic infusion. Patients allocated in the LBBAP group will be evaluated after the procedure and classified as LBBP or LVSP upon the accomplishment of the accepted criteria for LBBAP (consensus).

Consecutive patients requiring permanent pacemaker implantation due to high degree AVB according to current guidelines will be evaluated for inclusion in the study. All patients need to fit all inclusion criteria and none of the exclusion criteria.

Location of the right ventricle pacing lead. Right ventricle apical pacing (RVAP): Capture of the RV by apex stimulation, generating a QRS with LBBB morphology and superior axis.

Left bundle branch pacing (LBBP): Capture of the LBB in one of its ramifications, generating a QRS with RBBB morphology and variable duration, which depends on the grade of impairment present in the more distal conduction system. The rapid activation of the LBB leads to a short left ventricle activation time (LVAT), less than 80 msec, or a long V6-V1 inter peak time (IPT), more than 44 msec. Several other criteria have been described in order to confirm the LBB capture21,22.

Left ventricle septal pacing (LVSP): Only left septal myocardium is captured, obtaining a variable QRS duration with a RBBB morphology in V1, which often are acceptable in terms of similarity with LBBP, but criteria for LBBP are not met.

Deep septal pacing (DSP): Only deep septal myocardium is captured, obtaining a variable QRS duration and morphology, without a RBBB morphology in V1.

Procedure work-flow

The study arm will be defined by randomization immediately before the implantation. Patients randomized to RVAP group will undergo a regular classical apex ventricular lead. Patients randomized to LBBAP will be implanted as follows:

An EP recording system displaying the 12-leads ECG and at least one channel with intracardiac signals will be used in all cases to allow appropriate measurements and to assess the LBBAP criteria accoding to the 2023 Consensus. The 3 required criteria will be: the QRS morphology in V1, the left ventricle activation time (LVAT) and the interpeak V6 to V1 time (IPT). Other measures will be taken at operators' discretion.

Of importance, LBBAP implantation procedure will be similar for all patients: the CSP lead will be implanted in the left bundle branch area with anatomical guidance. Unipolar stimulation aiming for a "W" pattern in V1 will be performed during septal maping. Operators then will screw the lead, aiming for a moderate drop in the impedance, representing a deep penetration into the septum, together with the conversion of the "W" pattern into a qR or rSR pattern in lead V1. The current of injury (COI) will be additionally used to guide the penetration of the lead.

The cornerstone of this study will be to accept the first location as the final location, as long as unipolar and bipolar thresholds are optimal, and the RBBB pattern in lead V1 remains. To ensure a balanced distribution between LBBP and LVSP, the first operator will not have access to any criteria measurement during the implant procedure, but the morphology in V1. In case of suboptimal thresholds or absence of a RBBB in V1, operator will proceed to implant de lead in a different position. After the procedure investigators will fulfill the Redcap database with all the banned EPRS measurements.

Data collection and data analyses Data will be loaded to an electronic CRF (Redcap) by a local authorized operator after the implantation procedure and during each control visit. Every participant center will have access only to their local patients. Only the PI will have access to all the patients. At the end of the recruitment, all the data will analyzed. Variables will be expressed as mean ± SD or number of cases and proportions according to the variable type (Continuous or discrete). Normality will be tested using the Shapiro-Wilk test. Paired T-test will be used to compare 12 months LVEF and LVEDD vs basal LVEF and LVEDD in each group, and for other continuous variables. Z-test will be used to compare discrete variables. KM analyses and Multivariate analyses searching for predictors will be performed. Statistical analysis will be performed using STATA® version 15.2 for windows (StataCorp LLC, Texas).

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or more.
2. Preserved or mild deteriorated LVEF (Simpson >40%) assessed by a recent (<1 month before implantation) transthoracic echocardiography.
3. Indication for pacing based on the presence of a high degree AVB, and consequently with an anticipated high burden of ventricular pacing (>80%).
4. Life expectancy of more than 12 months and capability to understand the protocol, signing informed consent form, and complying with follow-up.

Exclusion Criteria:

1. Patients with indication for implantable cardioverter defibrillator device.
2. Patients with indication for a CRT device, with LVEF <40%.
3. Patients with previous severe LVD (Simpson LVEF <30%) and a recovered LVEF.
4. History of myocardial infarction/revascularization or cardiac surgery within 6 months before randomization.
5. Pregnancy, active cancer treatment, or participation in another clinical trial with active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
LVEF evolution | At 12 months after the pacemaker implantation
  Change in the value (%) of LVEF at 12 months compared to basal
Admission due to HF | From date of implantation until the date of first admission due to HF, whichever came first, assessed up to 12 months
  Hospital admission due to episode of heart failure (new onset HF or worsening from baseline NYHA)

SECONDARY OUTCOMES:
LVEED evolution | At 12 months after the pacemaker implantation
  Change in left ventricle end dyastolic diametre from the baseline, at 12 months from pacemaker implantation
Admission due to AF | From date of implantation until the date of first admission due to AF, whichever came first, assessed up to 12 months
  Hospital admission due to atrial fibrillation (new onset or relapse) after the pacemaker implantation

OTHER OUTCOMES:
Change in ProBNP | At 12 months after the pacemaker implantation
  Change in the value of pro-BNP at 12 months compared to baseline before pacemaker implantation
NYHA evolution | At 12 months after the pacemaker implantation
  Change in the NYHA heart failure class at 12 months compared to baseline
MLWHFQ evolution | At 12 months after the pacemaker implantation
  Change in the Minessota Living With Heart Failure Questionnare at 12 months compared to baseline (0-105 points, being 105 de worse situation)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar - IMIM, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD can be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD can be available in January of 2027, until January of 2037
Access Criteria: IPD will be available to any investigator request if the proposal is satisfatory

REFERENCES:
- [Background] Gonzalez-Matos CE, Rodriguez-Queralto O, Zaraket F, Jimenez J, Casteigt B, Valles E. Conduction System Stimulation to Avoid Left Ventricle Dysfunction. Circ Arrhythm Electrophysiol. 2024 Feb;17(2):e012473. doi: 10.1161/CIRCEP.123.012473. Epub 2024 Jan 29. PMID 38284238